CLINICAL TRIAL: NCT04891263
Title: Safety and Efficacy of Suture-Septoplasty for Chronic, Durable Correction of Nasal Septal Deviation Causing Nasal Obstruction Symptoms
Brief Title: Suture-based, Minimally Invasive Technique Used to Correct NSD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment difficulties due to COVID-19 pandemic
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Jayakar Nayak, Associate Professor of Otolaryngology - Head & Neck Surgery (OHNS) and, by courtesy, of Neurosurgery at the Stanford University Medical Center, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 57545
Record Dates: First submitted 2021-05-13; First posted 2021-05-18 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Nasal Septum; Deviation, Congenital; Nasal Obstruction
Keywords: septoplasty; suture-septoplasty; excisional septoplasty
MeSH Terms: conditions — Nasal Obstruction | interventions — Sutures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Suture-Septoplasty (Experimental): Participants will receive suture-septoplasty technique, and will be followed for three months postoperatively.
  Interventions: Procedure: Suture-Septoplasty; Device: Surgical suture

INTERVENTIONS:
Procedure: Suture-Septoplasty — Patients receive suture-septoplasty for repair of nasal septal deviation.
Device: Surgical suture — Suture used for closure during septoplasty surgery.
  Other Names: PDS suture

SUMMARY:
Nasal Septal Deviation (NSD) is one of the most common indications for surgery seen by ENT physicians, however, correction requires open surgery which is associated with several weeks of recovery. The purpose of this study is to elucidate whether a suture-based, minimally invasive technique can be used to safely and effectively address NSD.

DETAILED DESCRIPTION:
Nasal obstruction due to structural issues such as nasal septal deviation (NSD) is remarkably common. NSD is caused by warping of the midline cartilage and bone of the septum, which starts between the 2 nostrils, and extends 7 cm posteriorly to the nasopharynx. This crooked or deviated conformation in the nasal septum cartilage and/or bone leads to physical blockade of normal airflow through the nose, often leading to complaints of nasal congestion, sleep disturbance, exercise limitations, and even poor compliance with CPAP mask use for treatment of obstructive sleep apnea (OSA). To correct this structural issue in symptomatic patients, septoplasty surgery under general anesthesia is typically advocated.

As an alternative to standard septoplasty, there are rare reports of simplified suture techniques that may be used to straighten the nasal septal cartilage. However, virtually all published studies to our knowledge have still required 1) some degree of cartilage/bone excision, which can destabilize the nasal support framework, and 2) use of non-locking sutures which can break, provide insufficient support, and be technically challenging given that it requires knot tying within the narrow nasal cavity corridors.

The investigators have demonstrated in benchtop models that similar results to standard septoplasty techniques can may be achieved with the use of a non-retractable suture without the need for cartilage excision. This technique, therefore, could allow for a simple, and knotless, minimally invasive way to improve and/or correct symptomatic NSD.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Patients from all ethnic and geographic backgrounds within the Stanford Sinus Center with symptomatic NSD
* Primary patients with NSD without past septum surgery
* Patients who have failed maximum medical therapy
* Patients whose symptoms, examination and/or imaging findings are sufficiently severe as to warrant septoplasty as determined by the treating surgeon

Exclusion Criteria:

* Age < 18
* Recent surgery of any kind (<1 month)
* Inpatients
* Previous nasal septum surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2021-08-02 (Actual); Primary Completion 2021-09-13 (Actual); Study Completion 2021-09-13 (Actual)

PRIMARY OUTCOMES:
Nasal Obstruction Symptom Evaluation (NOSE) score | baseline, month 3
  Unabbreviated scale title: Nasal Obstruction Symptom Evaluation. Mean change from baseline. Minimum value = 0, maximum value = 100. Higher score indicates a worse outcome.

SECONDARY OUTCOMES:
Sino-Nasal Outcome Test (SNOT)-22 score | baseline, month 3
  Unabbreviated scale title: Sino-Nasal Outcome Test. Mean change from baseline. Minimum value = 0, maximum value = 110. Higher score indicates a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Jayakar V Nayak, M.D., Ph.D., Principal Investigator — Associate Professor of Otolaryngology - Head & Neck Surgery, Stanford University Medical Center
Locations (2):
- United States (2):
  - Stanford Ambulatory Surgery Center, Stanford Hospital, Palo Alto, California
  - Stanford Sinus Center/ Adult Comprehensive ENT Clinic, Stanford, California

IPD SHARING:
Plan to Share IPD: No
Only research personal listed in the IRB will have full access to PHI upon approval of the protocol director. All other participants conducting research pertaining to this study will receive anonymous information related to patient outcome that will not be linked to a patient identifier (including participant ID numbers).

REFERENCES:
- [Background] van Egmond MMHT, Rovers MM, Hannink G, Hendriks CTM, van Heerbeek N. Septoplasty with or without concurrent turbinate surgery versus non-surgical management for nasal obstruction in adults with a deviated septum: a pragmatic, randomised controlled trial. Lancet. 2019 Jul 27;394(10195):314-321. doi: 10.1016/S0140-6736(19)30354-X. Epub 2019 Jun 18. PMID 31227374
- [Background] Tan KH. Long-term survey of prominent ear surgery: a comparison of two methods. Br J Plast Surg. 1986 Apr;39(2):270-3. doi: 10.1016/0007-1226(86)90100-1. PMID 3697576
- [Background] Rigg BM. Suture materials in otoplasty. Plast Reconstr Surg. 1979 Mar;63(3):409-10. doi: 10.1097/00006534-197903000-00022. PMID 154115
- [Background] Boenisch M, Mink A. Clinical and histological results of septoplasty with a resorbable implant. Arch Otolaryngol Head Neck Surg. 2000 Nov;126(11):1373-7. doi: 10.1001/archotol.126.11.1373. PMID 11074836
- [Background] Gruber RP, Nahai F, Bogdan MA, Friedman GD. Changing the convexity and concavity of nasal cartilages and cartilage grafts with horizontal mattress sutures: part I. Experimental results. Plast Reconstr Surg. 2005 Feb;115(2):589-94. doi: 10.1097/01.prs.0000150145.39509.db. PMID 15692369
- [Background] Gruber RP, Nahai F, Bogdan MA, Friedman GD. Changing the convexity and concavity of nasal cartilages and cartilage grafts with horizontal mattress sutures: part II. Clinical results. Plast Reconstr Surg. 2005 Feb;115(2):595-606; discussion 607-8. doi: 10.1097/01.prs.0000150146.04465.81. PMID 15692370
- [Background] Seo HJ, Denadai R, Vamvanij N, Chinpaisarn C, Lo LJ. Primary Rhinoplasty Does Not Interfere with Nasal Growth: A Long-Term Three-Dimensional Morphometric Outcome Study in Patients with Unilateral Cleft. Plast Reconstr Surg. 2020 May;145(5):1223-1236. doi: 10.1097/PRS.0000000000006744. PMID 32332542
- [Background] Rohrich RJ, Friedman RM, Liland DL. Comparison of otoplasty techniques in the rabbit model. Ann Plast Surg. 1995 Jan;34(1):43-7. doi: 10.1097/00000637-199501000-00009. PMID 7702300
- [Background] Boenisch M, Tamas H, Nolst Trenite GJ. Influence of polydioxanone foil on growing septal cartilage after surgery in an animal model: new aspects of cartilage healing and regeneration (preliminary results). Arch Facial Plast Surg. 2003 Jul-Aug;5(4):316-9. doi: 10.1001/archfaci.5.4.316. PMID 12873869